CLINICAL TRIAL: NCT00608439
Title: Centella Asiatica Triterpene Extract for Diabetic Neuropathy -- a Pilot Study
Brief Title: Centella Asiatica Selected Triterpenes (CAST) for Diabetic Neuropathy
Acronym: CAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Jau-Shin Lou, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT003668 (NIH); R21AT003668 (NIH)
Record Dates: First submitted 2008-01-28; First posted 2008-02-06 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Diabetic Neuropathy
Keywords: CAST; Centella asiatica; Diabetes; Diabetic neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus | interventions — Centella asiatica extract; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo CAST
  Interventions: Drug: Centella asiatica selected triterpenes (CAST)
- Centella asiatica selected triterpenes (Active Comparator): Active CAST
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Centella asiatica selected triterpenes (CAST) — Drug provided to subjects in 60 mg capsules. Dose escalation phase: subjects take 2 capsules/day for weeks 1-4, 3 capsules/day for weeks 4-8 and 4 capsules/day weeks 8-12. Subjects remain on highest tolerated dose from week 12 to 52.
  Other Names: Centella asiatica; Gotu Kola
  Arms: Placebo
Other: Placebo — Placebo provided to subjects in 60 mg color-matched capsules. Dose escalation phase: subjects take 2 capsules/day for weeks 1-4, 3 capsules/day for weeks 4-8 and 4 capsules/day weeks 8-12. Subjects remain on highest tolerated "dose" from week 12 to 52.
  Other Names: Sugar pill
  Arms: Centella asiatica selected triterpenes

SUMMARY:
The purpose of this protocol is to investigate the safety, tolerability and effectiveness of CAST as a treatment for diabetic neuropathy. The primary outcome measure will be Total Neuropathic Symptom Score. Secondary outcomes will be neurological disability score, nerve conduction measurements and quantitative sensory testing. Statistical analyses will compare changes from baseline for CAST- and placebo-treated groups at both time points, compare effects of CAST at 6 and 12 months and, if numbers permit, compare doses.

DETAILED DESCRIPTION:
This study is a clinical trial investigating the effect of an herbal supplement called CAST on diabetic neuropathy. CAST is an herb commonly used in traditional Indian medicine. In this tradition, it is used to increase memory, treat wounds and sores, skin diseases, and neurological conditions such as epilepsy. The herb has had growing popularity in the US; parts are sold as the dietary supplement "gotu kola" and used to improve blood circulation and help heal wounds. Unlike many other herbs, CAST has been extensively researched for many of the above conditions. The compounds found in CAST make it a very promising potential treatment for diabetic neuropathy because of its effect on blood circulation and growth of nerves.

Subjects will receive informed consent. They will then be screened for eligibility before entering the study. A medical history will be taken and subjects will have a neurological exam and vital signs taken. Subjects will have their blood drawn and will also give a urine sample for routine testing. Subjects will have an electrocardiogram (ECG) to check their heart. If a subject is a woman who is at risk of getting pregnant, she will have a urine pregnancy test.

If the subject is eligible for participation in the study, they will return for a total of nine additional study visits over the course of a year. Subjects will be randomly assigned to either receive the active supplement (CAST) or a placebo. A placebo is a pill that tastes, looks, and smells like the study drug but has no real medicine (or supplement) in it. Subjects have a 50% chance of receiving the active supplement. Neither the subject nor the study staff will know who receives the active supplement or the placebo. At visits 2, 7 and 10, subjects will get a comprehensive assessment of their neuropathy symptoms. This will include a Neurological Disability Score assessment, a nerve conduction study and a Quantitative Sensory Test.

Subjects enrolled in the study will begin taking their study pills at the beginning of week 1 of the study. During the first 12 weeks, subjects will be asked to increase their dose by one pill every four weeks. Therefore, they will increase the number of CAST or placebo pills from 60mg twice daily to 60mg four times daily, or the highest dose that does not cause side effects. Dr. Lou will monitor subjects for side effects of the study supplement. At each study visit, blood and urine samples will be taken for safety analysis, including liver and kidney function, and glucose control, and an ECG will be done to monitor heart activity. Subjects will be contacted by the study coordinator via phone call once per week during the first three months of the study. During the remainder of the study, they will be called once each month that they are not scheduled for an appointment. Treatment will conclude after one year.

ELIGIBILITY:
Inclusion Criteria:

1. Type II diabetes that is being treated with diet, oral antidiabetic agents and/or insulin
2. stable glycemic control over the last 3 months
3. evidence of symptomatic symmetrical distal neuropathy
4. total symptom score of 4 or more
5. stable HbA1c level of less than 8.5 over last three months

Exclusion Criteria:

1. Smokers
2. Asymmetrical neuropathy of the trunk and proximal lower limbs
3. Presence of foot ulcers
4. Peripheral vascular disease (non-palpable foot pulses, intermittent claudication)
5. Myopathy
6. Causes of neuropathy other than diabetes
7. Participation in a study of any investigational drug for diabetic neuropathy within 3 months of the study
8. Use of any other product containing CA in the last 3 months
9. Starting to use antioxidants or Vitamin B within 1 month before the study
10. Severe concomitant diseases including neurological disease
11. Pregnancy, lactation or being of child-bearing age without birth control
12. HBA1c level higher than 8.5
13. Use of any experimental drugs in the three months prior to start of the study
14. Use of anti-coagulant therapy (heparin or coumarin based drugs)
15. A QTc of more than 500 ms at baseline ECG
16. Uncontrollable hypertension, defined as diastolic pressure greater than 110, and systolic pressure greater than 160

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Total Symptom Score | one year

SECONDARY OUTCOMES:
Nerve Conduction Study | one year
Neurological Disability Test | one year
Quantitative Sensory Test | one year

CONTACTS AND LOCATIONS:
Overall Officials: Jau-Shin Lou, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States